CLINICAL TRIAL: NCT04932590
Title: Predicting Fluid Responsiveness During Shock State by End-expiratory Occlusion Test in Newborns and Infants : EVEOC Study
Brief Title: Predicting Fluid Responsiveness During Shock in Newborns and Infants by End-expiratory Occlusion Test
Acronym: EVEOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP201320; ID RCB 2020-A02 (Other: ID-RCB Number)
Record Dates: First submitted 2021-06-14; First posted 2021-06-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Shock
Keywords: Shock; Invasive mechanical ventilation; Fluid responsiveness; Heart-lung interactions; End-expiratory occlusion test; Newborns and infants
MeSH Terms: conditions — Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental): Patients less than 2 years old admitted in the pediatric intensive care unit of the Armand-Trousseau hospital, under invasive mechanical ventilation and in whom a volume expansion is planned by the attending physicians.
  Interventions: Other: End-expiratory occlusion test

INTERVENTIONS:
Other: End-expiratory occlusion test — The test consists in interrupting the ventilator at end-expiration for 15 seconds and assessing the resulting changes in cardiac output. Delays necessary to allow sufficient pulmonary transit time to allow good pulmonary venous return and therefore an increase in cardiac preload.

SUMMARY:
To date, the end-expiratory occlusion test in infants or children has never been evaluated as a marker of preload dependence. It therefore appears clinically relevant to evaluate this new indicator to predict fluid responsiveness in all infants hospitalized in pediatric and neonatal intensive care.

The main objective of this study is to determine whether the hemodynamic effects of a 15-second end-expiratory occlusion were able to predict fluid responsiveness in the mechanically ventilated infant or newborn in pediatric intensive care.

DETAILED DESCRIPTION:
Volume expansion remains one of the first resuscitation treatments for states of shock. Nonetheless, the decision to perform volume expansion should be based on a "functional" hemodynamic assessment, i.e., filling should only be performed if changes in cardiac preload result in significant changes in stroke volume. This is then referred to as preload dependency. Unnecessary volume expansion induces fluid overload and is associated with increased morbidity and mortality for shock conditions in infant and children.

In addition, several studies in adults and children have demonstrated the lack of effectiveness of so-called "static" preload variables as witnesses of preload dependence. Only "dynamic" preload variables, based on the notion of cardiopulmonary interaction during mechanical ventilation, can predict this preload dependence, however with very variable sensitivities and specificities depending on the studies.

The end-expiratory occlusion test is a dynamic preload dependency test that can be performed in patients on invasive ventilation. The test consists in interrupting the ventilator at end-expiration for 15 seconds, delaying the next insufflation thus allowing an increase in venous return to the right heart and then to the left heart. If the heart is preload dependent, an increase in venous return is accompanied by an increase in stroke volume and cardiac output (Franck-Starling's law). Volume expansion is usually considered effective or positive if cardiac output increases by more than 15% from baseline.

To date, the end-expiratory occlusion test in infants or children has never been evaluated as a marker of preload dependence. It therefore appears clinically relevant to evaluate this new indicator to predict fluid responsiveness in all infants hospitalized in pediatric and neonatal intensive care.

The main objective of this study is to determine whether the hemodynamic effects of a 15-second end-expiratory occlusion were able to predict fluid responsiveness in the mechanically ventilated infant or newborn in pediatric intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Newborn and infant <2 years.
* Born at or near term (> 36 weeks of amenorrhea).
* Hospitalized in pediatric and neonatal intensive care.
* Requiring the use of invasive mechanical ventilation.
* In a state of shock defined by a cardio-circulatory dysfunction associating arterial hypotension, an alteration in organ perfusion, one or more organ dysfunctions or vasopressor's requirement. Clinical signs retained: heart rate ≥ 90th percentile associated with at least one sign of peripheral hypoperfusion represented by a a capillary refill time ≥ 3sec, or the presence of mottling or coldness of the extremities or urine output ≤ 0.5ml / kg / h or disturbance of consciousness.
* The practitioner in charge of the patient has decided to perform volume expansion.
* Non-opposition expressed by the holders of parental authority.

Exclusion Criteria:

* Any serious and urgent clinical hemodynamic situation, the management of which would be delayed by inclusion in the protocol.
* Patient with unoperated congenital heart disease.
* Patient in spontaneous or non-invasive ventilation or with spontaneous ventilatory cycles in invasive ventilation.
* Patient in prolonged cardiac arrest (> 5min) or refractory.
* Patient under venous-arterial extracorporeal membrane oxygenation.
* Refusal of the holders of parental authority to exploit the collected data.

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2021-12-24 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Cardiac output | 25 minutes
  Cardiac output measured by cardiac ultrasound before and during end-expiratory occlusion and after volume expansion.
  A positive response to end-expiratory occlusion is defined as an increase in cardiac output ≥ 15%.
  A positive response to the volume expansion test is defined as an increase in cardiac output ≥ 15%.

SECONDARY OUTCOMES:
Heart rate | 25 minutes
  Heart rate measured by cardiac ultrasound before and during end-expiratory pause and after volume expansion.
Systolic and diastolic blood pressures and mean arterial pressure | 25 minutes
  Recorded using a bedside monitor before and during end-expiratory pause and after volume expansion.
Arterial pulse pressure | 25 minutes
  Pressure waveform analysis was performed online with the soft tracing provided by the monitor.
  ∆PP (%) = PP max-PP min)/[(PP max+PP min)/2] × 100).
Stroke volume | 25 minutes
  Measured by cardiac ultrasound before and during end-expiratory pause and after volume expansion.
Aortic velocity time integral | 25 minutes
  Measured by cardiac ultrasound before and during end-expiratory pause and after volume expansion.
Aortic blood flow velocity | 25 minutes
  Measured by cardiac ultrasound before and during end-expiratory pause and after volume expansion.

CONTACTS AND LOCATIONS:
Overall Officials: Yaël LEVY, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Pierre-Louis LEGER, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Armand Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: No